CLINICAL TRIAL: NCT06251765
Title: Clinical Results After Judet Quadricepsplasty for Post-traumatic Knee Stiffness: a Retrospective and Prospective Observational Study
Brief Title: Clinical Results After Judet Quadricepsplasty for Post-traumatic Knee Stiffness
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: JUD-TR
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Knee Fractures; Stiffness of Knee, Not Elsewhere Classified
Keywords: arthromyolisis; Judet; post-traumatic; quadricepsplasty
MeSH Terms: conditions — Knee Fractures | interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who underwent Judet arthromyilisis for treatment of post-traumatic knee stiffness
  Interventions: Other: Clinical scores; Other: Range of Motion

INTERVENTIONS:
Other: Clinical scores — Clinical scores will be administered to patients
Other: Range of Motion — Evalutation of knee mobility

SUMMARY:
The Post-traumatic Extension Contracture of the Knee (PECK) is a common complication following knee traumas. It is characterized by a restricted Range of Motion (ROM), pain, and discomfort in the affected knee.

Various factors can cause PECK, primarily inflammation and scar tissue formation. The underlying inflammatory state leads to the development of scar tissue, which - when combined with immobilization - results in the progressive stiffness of the knee. Additionally, prolonged immobilization leads to muscle atrophy and, consequently, reduced mobility and increased rigidity.

All these conditions contribute to a limited ROM, making it challenging to perform various daily activities.

Sometimes conservative treatments can be effective, but surgery is often necessary to restore joint functionality and alleviate pain.

Historically, various surgical approaches have been proposed to address post-traumatic knee stiffness.

Open surgery is typically reserved for cases where arthroscopic adhesion release and manipulation under anesthesia have not been successful. Over the last century, various open surgical techniques have been proposed.

In particular, arthromyolysis according to Judet was first described in the 1950s by the French orthopedic surgeon Jacques Judet. This technique involves a series of incisions and soft tissue releases, allowing the surgeon to resolve the stiffness of the quadriceps tendon caused by trauma or prolonged immobilization.

Although effective in restoring knee joint functionality, arthromyolysis according to Judet is not without risks and potential complications. These include infection, massive bleeding, nerve and muscle-tendon injuries, and residual stiffness.

The purpose of this study is to analyze our case series related to arthromyolysis according to Judet for PECK. Clinical outcomes, complications, and patient satisfaction following this type of intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients underwent surgical intervention for arthromyolysis according to Judet with modified surgical technique for knee stiffness from January 2008 to December 2019.
2. Patients with post-traumatic injuries (fractures treated surgically).
3. Patients with a minimum of 4 years of follow-up.
4. Completeness of clinical documentation.

Exclusion Criteria:

1. Patients who underwent surgical intervention for arthrolysis (both arthroscopic and non-arthroscopic) or arthromyolysis according to Judet with minimally invasive technique.
2. Patients who underwent surgery to address knee stiffness due to other causes (rigid prosthesis, limb lengthening, etc.).
3. Incomplete clinical documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent Judet arthromyolisis for treatment of post-traumatic knee-stiffness
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Range of Motion at follow-up | baseline time 0
  ROM expresses in degrees the degree of range of motion that a joint can perform along its full range of motion whether active or passive through an external aid.

SECONDARY OUTCOMES:
Intra-operative Range of Motion | baseline time 0
  ROM expresses in degrees the degree of range of motion that a joint can perform along its full range of motion whether active or passive through an external aid.
Knee injury and Osteoarthritis Outcome Score | baseline time 0
  KOOS assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Tegner Activity Scale | baseline time 0
  Tegner Activity Scale is used in order to provide a standardized method to grade work and sporting activities.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pujol N, Boisrenoult P, Beaufils P. Post-traumatic knee stiffness: surgical techniques. Orthop Traumatol Surg Res. 2015 Feb;101(1 Suppl):S179-86. doi: 10.1016/j.otsr.2014.06.026. Epub 2015 Jan 9. PMID 25583236
- [Result] Luo Y, Li H, Mei L, Mao X. Effects of Judet Quadricepsplasty in the Treatment of Post-traumatic Extension Contracture of the Knee. Orthop Surg. 2021 Jun;13(4):1284-1289. doi: 10.1111/os.12950. Epub 2021 May 6. PMID 33955701
- [Result] Bidolegui F, Pereira SP, Pires RE. Safety and efficacy of the modified Judet quadricepsplasty in patients with post-traumatic knee stiffness. Eur J Orthop Surg Traumatol. 2021 Apr;31(3):549-555. doi: 10.1007/s00590-020-02802-3. Epub 2020 Oct 13. PMID 33051692